CLINICAL TRIAL: NCT05014633
Title: The Effect of Training on the Promotion of Emotional Intelligence and Its Indirect Role in Reducing Job Stress in the Emergency Department
Brief Title: The Effect of Emotional Intelligence in Reducing Job Stress
Acronym: EI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Principal Investigator, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 960235
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Emotional Intelligence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EI skills training (Experimental): Individuals in the intervention group received the pertinent training. The duration of the training for the intervention group was 16 hours (four four-hour sessions). The whole training process lasted for one month. EI training sessions were held and managed by two experienced instructors selected from medical education specialists with sufficient experience in conducting EI training. Both instructors attended the sessions, presented the content, videos, slides, and brochures with the help of each other, and managed related scenarios in each session.
  Interventions: Other: EI skills training
- Control (No Intervention): Individuals in the control group did not receive any training

INTERVENTIONS:
Other: EI skills training — EI training sessions were held and managed by two experienced instructors selected from medical education specialists with sufficient experience in conducting EI training. Both instructors attended the sessions, presented the content, videos, slides, and brochures with the help of each other, and managed related scenarios in each session.
  Arms: EI skills training

SUMMARY:
Abstract Background: Emergency Medicine Wards (EMWs) are among the most stressful wards of hospitals. Emotional Intelligence (EI) seems to be one of the factors that can aid individuals in overcoming environmental stresses. Therefore, the present study aimed at evaluating the role of training in improving EI skills and addressing its indirect effect on reducing job stress of emergency medical assistants in the emergency department.

Materials and Methods: In the present study, 20 emergency medical assistants were trained in EI skills while 22 assistants received no training. Then, all participants' EI level and job stress were assessed and compared before and after the intervention using the Bar-On Emotional Quotient Inventory(EQ-i) and the Osipow job stress questionnaire, respectively.

DETAILED DESCRIPTION:
Individuals in the control group did not receive any training while individuals in the intervention group received the pertinent training. The duration of the training for the intervention group was 16 hours (four four-hour sessions). The whole training process lasted for one month. EI training sessions were held and managed by two experienced instructors selected from medical education specialists with sufficient experience in conducting EI training. Both instructors attended the sessions, presented the content, videos, slides, and brochures with the help of each other, and managed related scenarios in each session.

It should be noted that the instructors as well as the participants had no information about the initial scores of EI and job stress recorded before the training intervention.

At the beginning of the first session, the basic definitions and concepts of EI were discussed, and the common environmental stressors were described from the perspective of emergency medical assistants. Moreover, a succinct description of the benefits of EI training and practice was provided. After the initial introduction, a number of EI skills were taught in each session by presenting videos, slides, and brochures. Then, participants were engaged in discussions by presenting scenarios related to EI skills in the concluding hours of each session to offer more content load. These scenarios recounted the situation of an individual facing a problem and encompassed a list of suggested reactions including the reasons behind each reaction that an observer was supposed to indicate. Scenarios were generally implemented in smaller groups in such a way that some scenarios were distributed and discussed among all participants. The assistants were questioned about identifying the source of the concern, the cause of the concern, potential environmental factors, and how a personal perspective affects their response to the situation. Other scenarios were distributed among the smaller groups and discussed by each groups' representative. Each group presented their analysis and argumentation of the scenario, and then the relevant questions were answered by providing the reasons. The sessions ended with the instructor summarizing different opinions on each of the scenarios (19).

It should be mentioned that to prevent fatigue and obtain better efficiency, participants (emergency medical assistants) were served twice during each session. Moreover, considering the possibility of the interference of emergency medical assistants' work shifts, it was planned in coordination with the Deputy Minister of Education that the emergency medical assistants would not have any work shifts and would not even be on duty over the four days of training.

Outcomes At the end of the last training session, two questionnaires of EQ-I and Osipow were filled out by the participants of the intervention group. In addition, the participants of the control group were contacted and asked to fill out these two questionnaires by visiting them in person (on the last day of the training session related to the intervention group). If the participant in the control group did not meet the conditions for the face-to-face visit, the questions were read to them on the phone and their choice was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine Residents

Exclusion Criteria:

* Refraining to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
EQ-I Bar-On Questionnaire | 30 days
  The EQ-I was first developed by Bar-On in 1980 and consists of 90 items, each of which is answered based on a 5-point Likert scale from 5: strongly agree to 1: strongly disagree

SECONDARY OUTCOMES:
Osipow job stress Questionnaire | 30 days
  The Osipow job stress questionnaire was first developed by Osipow and Spokane in 1987 and consists of 60 items, each of which is answered based on a 5-point Likert scale from 4: most of the time to 0: never.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Nasr Isfahani, M.D., Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Al-Zahra University Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No